CLINICAL TRIAL: NCT04696588
Title: Physiotherapy Methods in Tinnitus Treatment
Brief Title: Neck Kinesiotherapy and Massage in Tinnitus Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESITESR14
Record Dates: First submitted 2019-12-10; First posted 2021-01-06 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Subjective Tinnitus
Keywords: Subjective tinnitus,; massage; Post Isometric Relaxation Exercises; Kinesiotherapy
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: It is a non randomized controlled trial
Who Masked: Investigator
Masking Description: The responsible investigator is blinded .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotherapy group (Experimental): This is the group (n=59) receives treatment i.e complex set of neck exercises and massage
  Interventions: Other: Complex set of kinesiotherapy of cervical spine and delicate massage
- Waiting List group (No Intervention): Individuals registered in the waiting list for receiving the treatment specified for kinesiotherapy group (n=59).These patients receive no treatment for tinnitus.

INTERVENTIONS:
Other: Complex set of kinesiotherapy of cervical spine and delicate massage — Intervention:- A complex neck therapy.Treatment comprises 10 sessions performed on consecutive working days, includes four parts.
  1. Active exercises of the neck, 5 minutes, first demonstrated by the physiotherapist and next the patient performs them under supervision, 5 repetitions of each of the following: cervical flexion, rotation to the left and to the right, side bending to the left and to the right, torsion to left and right.
  2. Massage of cervical interspinales muscles performed by therapist 3 minutes.
  3. Post Isometric Relaxation (PIR) performed by physiotherapist. 15 minutes.
  4. Active neck exercises - the same as mentioned in step 1. 5 minutes. Total duration of one treatment session is around 30 minutes.
  Arms: Kinesiotherapy group

SUMMARY:
The primary aim of this study is to investigate the effectiveness of cervical spine kinesiotherapy and massage in tinnitus treatment. Furthermore, we investigate if there is a link between cervical spine range of motion and cervical muscles tension and tinnitus.

DETAILED DESCRIPTION:
The study is planned with power of 80%. A total of 118 adult patients with subjective tinnitus are divided into two groups: Kinesiotherapy group (n=59) and Waiting list group (n=59).Kinesiotherapy group receives a complex set of cervical spine exercises and neck massage for consecutive 10 working days (entire treatment takes two weeks). Each visit lasts around 30 minutes. Patients from kinesiotherapy group will fill the outcome measures on the following time points: (a) Time point 0 - baseline (b) Time point 1- Two weeks after the baseline

(c) Time point 2- Four weeks after the baseline. Individuals from waiting list group are enrolled on a waiting list and do not receive any treatment. They undergo assessment at three time points corresponding to Kinesiotherapy group i.e Time point 0, Time point 1 and Time point 2.

.

ELIGIBILITY:
Inclusion Criteria:

-Adult patients with subjective tinnitus experienced in the ears or in the head (temporary and constant tinnitus) with and without sensorineural hearing loss.

Exclusion Criteria:

* Other tinnitus treatment in last 6 months,
* Objective tinnitus,
* External and middle ear pathology,
* Acute infections, conditions with fever
* Bleedings or risk of bleeding
* Severe respiratory and circulatory insufficiency
* vasculitis, thrombophlebitis,
* Pregnancy
* Acute arthritis and periarticular soft tissues inflammation in the cervical region,
* Severe pains in different locations,
* Advanced osteoporosis
* Uniformed services.
* Cervical spine instability, cervical disc herniation, cervical radiculopathy.
* Status post cervical spine surgery.
* Status post lumbar puncture, status post computed tomography with contrast.
* Lack of cooperation between the patient and the therapist, cognitive impairment.
* Atherosclerosis, vertebrobasilar insufficiency.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Tinnitus Functional Index (TFI), a Polish validated version (Wrzosek et al., 2016). | Time point 0: Baseline, Time point 1: 2 weeks after baseline, Time point 2: 4 weeks after baseline
  The Tinnitus Functional Index is a comprehensive scale, assessing tinnitus severity, comprising 25 questions. It has eight subscales: intrusiveness, sense of control, cognitive, sleep, auditory, relaxation, quality of life, and emotion. Patients can mark their response on a scale starting from zero (0) to maximum response (10). Maximum possible score of TFI is 250 if the respondent were to mark all 25 TFI items at the maximum value of 10. High scores on TFI scale are interpreted as increased severity of tinnitus and negative impact on patients life.
  Total TFI score is analyzed at three time points as described above. Statistical analysis is performed using repeated measures ANOVA to evaluate if there is a significant difference in the mean TFI score at the three time points.

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory (THI), Polish validated version | as for TFI
  2. Tinnitus Handicap Inventory (THI), Polish validated version
  Tinnitus Handicap Inventory measures the impact of tinnitus on the daily life of the patients. The questionnaire is subdivided into categories functional (11 questions), emotional (9 questions) and catastrophic (5 questions) :Tinnitus Handicap Inventory comprises 25 questions with three options for answer: "Yes", "NO", "Sometimes". The scoring for these options is "Yes"= 4,"NO "=0 ,"sometimes"=2. The possible score for Tinnitus Handicap Inventory can range from 0 to 100. Higher scores are interpreted as greater handicap due to tinnitus.Total THI score will be analyzed at three time points as for TFI.
Visual Analogue Scale (VAS) | as for TFI
  The Visual Analogue Scale (was used to asses subjective tinnitus loudness). The patient will report averaged loudness of their tinnitus in the past week on a 10 centimeter line. The left end of the line was marked with 0 indicating no tinnitus, while the right end was marked with 10, indicating maximum loudness of tinnitus. Visual Analogue scale score will be assessed on three time points - as for TFI. Visual Analogue scale score will be assessed on three time points - as for TFI.
Range of motion of cervical spine | as for TFI
  This is the range of neck movements that the patient can actively perform, measured from the neutral to maximum position (cervical flexion, cervical rotation to left and to right, cervical side bending to left and right. The SFTR method where S represents - sagittal (sagittal plane);
  - Page 3 of 6 [DRAFT] -
  F - Frontal plane; T - transverse (transverse plane); R - rotation (rotational movements) will be used for assessment and recording cervical spine range of movement (Gerhardt,1983). The normal range of movement of cervical spine according to SFTR method in centimetres, is as follows:
  Cervical Spine flexion
  * 18-40 years adults- 3 cm.
  * 41-60 years adults- 2.5 cm.
  * 61-85 years adults- 2 cm
  Cervical Side bending
  * 18-40 years adults- 6.5 cm.
  * 41-60 years adults- 5 cm.
  * 61-85 years adults- 4 cm
  Cervical rotation
  * 18-40 years adults- 8 cm.
  * 41-60 years adults- 7.5 cm.
  * 61-85 years adults- 6 cm.
Cervical muscle tension (MST) | same as for TFI
  The cervical muscle tension will be assessed by palpation. Palpation is widely used as a physiotherapy assessment tool in patient examination (MAITLAND, 1982). Muscle tension will be graded using the dichotomous scale of 0 and 1 where 0 will be interpreted as normal and 1 will be interpreted as presence of pathological muscle tension.

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Marzena Mielczarek, MD PhD, Principal Investigator — Medical University of Lodz Poland
Locations (1):
- Department of Otolaryngology, Laryngological Oncology, Audiology and Phoniatrics, Teaching Hospital of Medical university of Lodz, Poland, Lodz, Lodz, Zeromskiego 113 Street, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Result] Cleland JA, Mintken PE, Carpenter K, Fritz JM, Glynn P, Whitman J, Childs JD. Examination of a clinical prediction rule to identify patients with neck pain likely to benefit from thoracic spine thrust manipulation and a general cervical range of motion exercise: multi-center randomized clinical trial. Phys Ther. 2010 Sep;90(9):1239-50. doi: 10.2522/ptj.20100123. Epub 2010 Jul 15. PMID 20634268
- [Result] Wrzosek M, Szymiec E, Klemens W, Kotylo P, Schlee W, Modrzynska M, Lang-Malecka A, Preis A, Bulla J. Polish Translation and Validation of the Tinnitus Handicap Inventory and the Tinnitus Functional Index. Front Psychol. 2016 Nov 29;7:1871. doi: 10.3389/fpsyg.2016.01871. eCollection 2016. PMID 27965609
- [Result] Michiels S, De Hertogh W, Truijen S, Van de Heyning P. Cervical spine dysfunctions in patients with chronic subjective tinnitus. Otol Neurotol. 2015 Apr;36(4):741-5. doi: 10.1097/MAO.0000000000000670. PMID 25415466
- [Result] Michiels S, Harrison S, Vesala M, Schlee W. The Presence of Physical Symptoms in Patients With Tinnitus: International Web-Based Survey. Interact J Med Res. 2019 Jul 30;8(3):e14519. doi: 10.2196/14519. PMID 31364603
- [Result] Latifpour DH, Grenner J, Sjodahl C. The effect of a new treatment based on somatosensory stimulation in a group of patients with somatically related tinnitus. Int Tinnitus J. 2009;15(1):94-9. PMID 19842352
- [Result] Sanchez TG, Rocha CB. Diagnosis and management of somatosensory tinnitus: review article. Clinics (Sao Paulo). 2011;66(6):1089-94. doi: 10.1590/s1807-59322011000600028. PMID 21808880
- [Result] Michiels S, Naessens S, Van de Heyning P, Braem M, Visscher CM, Gilles A, De Hertogh W. The Effect of Physical Therapy Treatment in Patients with Subjective Tinnitus: A Systematic Review. Front Neurosci. 2016 Nov 29;10:545. doi: 10.3389/fnins.2016.00545. eCollection 2016. PMID 27965530
- [Result] Maitland GD. Palpation examination of the posterior cervical spine: the ideal, average and abnormal. Aust J Physiother. 1982 Jun;28(3):3-12. doi: 10.1016/S0004-9514(14)60768-6. PMID 25025844
- [Result] Gerhardt JJ. Clinical measurements of joint motion and position in the neutral-zero method and SFTR recording: basic principles. Int Rehabil Med. 1983;5(4):161-4. doi: 10.3109/03790798309167039. PMID 6662609